CLINICAL TRIAL: NCT02203526
Title: Phase 1 Study of Ibrutinib and Immuno-Chemotherapy Using Temozolomide, Etoposide, Doxil, Dexamethasone, Ibrutinib, Rituximab (TEDDI-R) in Primary CNS Lymphoma
Brief Title: Phase 1 Study of Ibrutinib and Immuno-Chemotherapy Using Temozolomide, Etoposide, Doxil, Dexamethasone, Ibrutinib,Rituximab (TEDDI-R) in Primary CNS Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 140157; 14-C-0157
Record Dates: First submitted 2014-07-29; First posted 2014-07-30 (Estimated); Last update posted 2026-01-28 (Actual); Status verified 2026-01-22

CONDITIONS: Primary Central Nervous System Lymphoma
Keywords: Tyrosine Kinase Inhibitor; ABC DLCBL; Lymphoma in Brain and CNS; Diffuse Large B-Cell Lymphomas in CNS
MeSH Terms: interventions — isavuconazole; Rituximab; Cytarabine; ibrutinib; Methotrexate

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Arm 1-A (original study design - prior to Amendment G) (Experimental): TEDD-R (cycle 1) with ibrutinib; TEDDI-R with cytarabine (cycles 2-6)
  Interventions: Drug: TEDDI; Biological: Rituximab; Drug: Cytarabine; Drug: TEDD; Drug: Ibrutinib (Arms 2, 3 and 4); Drug: Ibrutinib (Arm 1 - Closed with Amendment G); Drug: Ibrutinib (Arm 4)
- Arm 1-B (original study design-prior to Amendment G) (Experimental): TEDDI-R with cytarabine
  Interventions: Drug: TEDDI; Biological: Rituximab; Drug: Cytarabine
- Arm 2 (Dose Escalation; prior to Amendment 06/04/2021) (Experimental): TEDDI-R with cytarabine, and isavuconazole
  Interventions: Drug: Isavuconazole; Drug: TEDDI; Biological: Rituximab; Drug: Cytarabine
- Arm 3 (Dose Expansion; prior to Amendment 06/04/2021) (Experimental): TEDDI-R with cytarabine and isavuconazole
  Interventions: Drug: Isavuconazole; Drug: TEDDI; Biological: Rituximab; Drug: Cytarabine
- Arm 4 (Dose Expansion; Amendment 06/04/21) (Experimental): TEDDI-R, cytarabine or methotrexate, isavuconazole, ibrutinib for 10 days
  Interventions: Drug: Isavuconazole; Drug: TEDDI; Biological: Rituximab; Drug: Cytarabine; Drug: Methotrexate; Drug: Ibrutinib (Arm 4)

INTERVENTIONS:
Drug: Isavuconazole — Isavuconazole to begin at least 3 days prior to ibrutinib and continue throughout chemotherapy (cycles 1-6)
  Arms: Arm 2 (Dose Escalation; prior to Amendment 06/04/2021); Arm 3 (Dose Expansion; prior to Amendment 06/04/2021); Arm 4 (Dose Expansion; Amendment 06/04/21)
Drug: TEDDI — Temozolomide, etoposide, doxil, dexamthasone, ibrutinib (TEDDI) given every 21 days for cycles 2-6 (Arm 1-A); given every 21 days for cycles 1-6 (Arms 1-B, 2, 3 and 4)
Biological: Rituximab — Rituximab (R) given with TEDD and TEDDI every 3 weeks for cycles 1-6 (all arms)
Drug: Cytarabine — Cytarabine given via Ommaya reservoir (IT therapy) on days 1 and day 5 of cycles 2-6 (all arms)
Drug: TEDD — Temozolomide, etoposide, doxil, dexamthasone, (TEDD) given on first cycle (Arm 1-A)
  Arms: Arm 1-A (original study design - prior to Amendment G)
Drug: Ibrutinib (Arms 2, 3 and 4) — Ibrutinib given on day -3 to day -1 on cycle 1 (Arms 2, 3 and 4)
  Arms: Arm 1-A (original study design - prior to Amendment G)
Drug: Methotrexate — Methotrexate on days 1 and day 5 of cycles 2-6 (Arm 4)
  Arms: Arm 4 (Dose Expansion; Amendment 06/04/21)
Drug: Ibrutinib (Arm 1 - Closed with Amendment G) — Ibrutinib given on day -14 to day -1 on cycle 1 (Arm 1)
  Arms: Arm 1-A (original study design - prior to Amendment G)
Drug: Ibrutinib (Arm 4) — Ibrutinib given on days 1-10 for cycles 1-6 (Arm 4)
  Arms: Arm 1-A (original study design - prior to Amendment G); Arm 4 (Dose Expansion; Amendment 06/04/21)

SUMMARY:
BACKGROUND:

* Primary CNS lymphoma (PCNSL) is a rare subtype of diffuse large B-cell lymphoma.
* The outcome for patients with this diagnosis is significantly worse than for that of systemic DLBCL. Most treatment approaches in the past have included high dose methotrexate and radiation treatment.
* Most PCNSLs appear to be of activated B-cell (ABC) origin.
* Ibrutinib is an inhibitor of Bruton s tyrosine kinase (BTK) and effective for systemic DLBCL of ABC origin.
* We propose doing a study in which ibrutinib is combined with a novel chemotherapy platform called dose adjusted temozolomide, etoposide, doxil, dexamethasone, ibrutinib, rituximab (TEDDI-R).

OBJECTIVE:

- Identify the maximum tolerated dose (MTD) of ibrutinib or the dose that achieves adequate CSF concentrations, whichever comes first, when ibrutinib is given with TEDDI-R.

ELIGIBILITY:

* Relapsed/refractory PCNSL.
* Age greater than or equal to 18 years.
* No pregnant or breast-feeding women.
* Adequate organ function (defined in protocol).

STUDY DESIGN:

* This is a phase 1 study of 40 patients.
* The study will have two components.

  1. Phase 1: MTD of ibrutinib will be identified or the dose at which ibrutinib achieves a concentration of less than or equal to 100 nM in the CSF, when given in combination with TEDDI-R immuno-chemotherapy, whichever comes first.
  2. Expansion cohort: Safety and tolerability of the regimen in relapsed/refractory or previously untreated PCNSL (DLBCL type) will be assessed at the final ibrutinib dose with TEDDI-R in 10 patients. Secondary objectives will be PFS and OS.

DETAILED DESCRIPTION:
Background:

* Primary CNS lymphoma (PCNSL) is a rare subtype of diffuse large B-cell lymphoma
* The outcome for patients with this diagnosis is significantly worse than for that of systemic DLBCL. Most treatment approaches in the past have included high dose methotrexate and radiation treatment.
* Most PCNSLs appear to be of activated B-cell (ABC) origin
* Ibrutinib is an inhibitor of Bruton's tyrosine kinase (BTK) and effective for systemic DLBCL of ABC origin.
* We propose doing a study in which ibrutinib is combined with a novel chemotherapy platform called temozolomide, etoposide, doxil, dexamethasone, ibrutinib, rituximab (TEDDI-R).

Objective:

* To identify the dose of ibrutinib with anti-fungal prophylaxis that can be safely administered to achieve an ibrutinib median CSF CMAX of 1.98 nM (Range 0.69 to 11.1)
* To assess the safety, feasibility, and complete response (CR) rate of the TEDDI-R in untreated PCNSL (DLBCL type) patients.

Eligibility:

* Relapsed/refractory or untreated PCNSL
* Age >= 18 years.
* No pregnant or nursing individuals.
* Adequate organ function (defined in protocol).

Study Design:

* This is a phase 1 study of 93 patients.
* The study will have three components.

  * Phase 1: MTD of ibrutinib will be identified or the dose at which ibrutinib achieves a concentration of >= 100 nM in the CSF, when given in combination with TEDDI-R immuno-chemotherapy, whichever comes first.
  * Expansion cohort: Safety and tolerability of the regimen in relapsed/refractory PCNSL (DLBCL type) will be assessed at the final ibrutinib dose with TEDDI-R in 10 patients. Secondary objectives will be PFS and OS.
  * Revised Study Design: new ibrutinib dose levels are being added together with anti-fungal prophylaxis to determine the dose of ibrutinib that may be safely given with the chemotherapy platform.
  * A second expansion cohort of untreated PCNSL (DLBCL type) will be added: Safety, feasibility, and complete response rate of the regimen in untreated PCNSL (DLBCL type) will be assessed at the final ibrutinib dose with TEDDI-R in 15 patients. Secondary objectives will be PFS and OS.
  * A new dosing schedule will be tested in up to 10 relapsed or refractory patients and 15 patients with untreated PCNSL. Secondary objectives will be PFS and OS.

ELIGIBILITY:
* ELIGIBILITY CRITERIA:
* Patients must have histologically or cytologically confirmed primary central nervous system diffuse large B-cell lymphoma. Patients with PCNSL that is only extracranial will not be eligible. Patients with relapsed or refractory disease, as well as untreated patients,

are eligible. Untreated patients must not have high dose chemotherapy and autologous stem cell transplantation (ASCT) planned as part of frontline therapy to be eligible for the trial.

* At least 2 weeks have passed since prior chemotherapy, biological therapy, radiation therapy, other investigational or anti-cancer therapy that is considered disease-directed.
* Ibrutinib must be discontinued 7 days before (when possible) until 7 days after major surgery, and 3 days before (when possible) until 3 days after minor surgery. Thus, patients to be enrolled on an ibrutinib trial must have completed major surgery >= 7 days before initiating treatment, and/or must have completed minor surgery >= 3 days before initiating treatment.
* Recovered from prior toxicities to Grade 0-1 at least 2 weeks prior to investigational therapy.
* Age >=18 years. Because no dosing or adverse event data are currently available on the use of ibrutinib and TEDDI-R in patients <18 years of age, children are excluded from this study, but may be eligible for future pediatric trials.
* ECOG performance status <=2 (Karnofsky >=60%) unless due to neurologic deficits caused by CNS lymphoma with the following exceptions: patients with ECOG PS = 4 where neurologic deficits are unlikely to resolve with tumor resolution and may cause clinical management problems are excluded.
* Patients must have normal organ and marrow function as defined below, independent of growth factor or transfusion support. Patients should not receive growth factors or transfusions for at least 7 days prior to first dose of study drug with the exception of pegylated G-CSF (pegfilgrastim) and darbepoeitin which require at least 14 days prior to screening and randomization.

  * absolute neutrophil count >= 750 cells/mcL (0.75 x 10(9)/L)
  * platelet count >= 50,000 cells/mcL (50 X 10(9)/L)
  * Hemoglobin > 8.0 g/dL
  * total bilirubin <=1.5 x ULN (unless Gilbert's syndrome or disease infiltration of the liver is present)
  * AST(SGOT)/ALT(SGPT) <= 3.0 x institutional ULN
  * Serum Creatinine <= 1.5 mg/dL OR creatinine clearance >= 40 ml/min/1.73m^2 unless lymphoma related.
* Prothrombin time/INR (PT) and activated partial thromboplastin time (aPTT) must be <= 1.5 x the upper limit of the normal range (ULN); except if, in the opinion of the Investigator, the aPTT is elevated because of a positive Lupus Anticoagulant.
* Left ventricular ejection fraction (LVEF) > 40% as assessed by echocardiogram
* The effects of ibrutinib on the developing human fetus are unknown. For this reason and because tyrosine kinase inhibitors as well as other therapeutic agents used in this trial may be teratogenic, individuals of reproductive potential and individuals who can father children must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry.
* Female patients who are of non-reproductive potential (i.e., post-menopausal by history - no menses for >=1 year; OR history of hysterectomy; OR history of bilateral tubal ligation; OR history of bilateral oophorectomy). Female patients of childbearing potential must have a negative serum pregnancy test upon study entry.
* Male and female patients must agree to use highly effective methods of birth control. A "highly effective method of birth control" is defined as a method that has a low failure rate (i.e., less than 1% per year) when used consistently and correctly and includes implants, injectables, birth control pills with two hormones, some intrauterine devices (IUDs). Male subject cannot use highly effective methods and are required to use barrier. The specific guidelines are as follows:

  * Individuals that bear children, must use a highly effective method of birth control and a barrier method, or sexual abstinence (which is defined as refraining from all aspects of sexual activity), while taking study treatment, as well as for 12 months after the last dose of rituximab.
  * Individuals who can father children must use a barrier method while on treatment with ibrutinib and for 3 months after the last dose of treatment to prevent pregnancy of your partner. Such individuals should donate sperm while you are taking the study drug and for 12 months after the last dose of rituximab.
* Patient or appointed surrogate decision-maker or legally authorized representative must have ability to understand the purpose and risks of the study and willingness to provide a signed and dated informed consent form (ICF) and authorization to use protected health information (in accordance with national and local subject privacy regulations).

EXCLUSION CRITERIA:

* Prior exposure to a BTK inhibitor.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ibrutinib or other agents used in study.
* Patients who are allergic to isavuconazole or any of its ingredients.
* Patients who received a strong cytochrome P450 (CYP) 3A inhibitor or inducer within 7 days prior to the first dose of protocol anti-fungal prophylaxis, or patients who require continuous treatment with a strong CYP3A inhibitor/inducer (i.e., with the exception of any medication to be specifically studied in this protocol).
* Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated list; medical reference texts such as the Physicians' Desk Reference may also provide this information. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product.
* HIV positive patients will be excluded because of their increased susceptibility to fungal infections which outweighs the potential benefit of participation.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or an infection requiring systemic antibiotics, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements. Recent infections requiring systemic treatment need to have completed therapy >14 days before the first dose of study drug.
* Pregnant and nursing individuals are excluded from this study. Pregnant individuals are excluded in this study because ibrutinib is a tyrosine kinase inhibitor with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of with a nursing participant ibrutinib, nursing should be discontinued if the mother is treated with ibrutinib.
* Uncontrolled Autoimmune Hemolytic Anemia or ITP resulting in (or as evidenced by) declining platelet or Hgb levels within the 4 weeks prior to first dose of study drug.
* Presence of transfusion-dependent thrombocytopenia.
* History of prior malignancy, with the exception of the following:

  * Malignancy treated with curative intent and with no evidence of active disease present for more than 3 years prior to Screening and felt to be at low risk for recurrence by treating physician
  * Adequately treated non-melanomatous skin cancer or lentigo maligna melanoma without current evidence of disease
  * Adequately treated carcinoma in situ without current evidence of disease.
* Currently active clinically significant cardiovascular disease such as uncontrolled arrhythmia, congestive heart failure, or Class 3 or 4 congestive heart failure as defined by the New York Heart Association Functional Classification, or history of myocardial infarction unstable angina, or acute coronary syndrome within 6 months prior to enrollment in the study.
* Unable to swallow capsules, or disease significantly affecting gastrointestinal function or resection of the stomach or small bowel, or symptomatic inflammatory bowel disease or ulcerative colitis, or partial or complete bowel obstruction.
* Serologic status reflecting active hepatitis B or C infection. Patients that are positive for hepatitis B core antibody, hepatitis B surface antigen (HBsAg), or hepatitis C antibody must have a negative polymerase chain reaction (PCR) prior to enrollment. Those who are PCR positive will be excluded. Those with a negative PCR for hepatitis B will be treated with antivirals designed to prevent hepatitis B reactivation (e.g., entecavir) and have monitoring for hepatitis B reactivation with PCR.
* History of stroke or intracranial hemorrhage within 6 months prior to enrollment.
* Any life-threatening illness, medical condition, or organ system dysfunction that, in the Investigator's opinion, could compromise the patient's safety, or put the study at undue risk. Patients with suspicious radiologic evidence of aspergillosis infection (i.e., Chest CT and/or Brain MRI) will not be eligible unless confirmatory laboratory testing of Beta-D glucan and aspergillus antigen are negative.
* Concomitant use of warfarin or other vitamin K antagonists within the last 7 days.
* Concurrent systemic immunosuppressant therapy other than corticosteroids (e.g., cyclosporine A, tacrolimus, etc.) within 28 days of the first dose of study drug.
* Vaccinated with live, attenuated vaccines within 4 weeks of first dose of study drug.
* Unresolved toxicities from prior anti-cancer therapy, defined as having not resolved to grade <=1, or to the levels dictated in the inclusion/exclusion criteria with the exception of alopecia.
* Known bleeding disorders (e.g., von Willebrand's disease) or hemophilia.
* Major surgery within 7 days of first dose of study drug.
* Unwilling or unable to participate in all required study evaluations and procedures.
* Currently active, clinically significant hepatic impairment (>= moderate hepatic impairment according to the NCI/Child Pugh classification)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Estimated)
Dates: Start 2014-08-14 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
safety and feasibility in untreated PCNSL patients | Initiation of ibrutinib until 30 days after treatment
  Incidence of adverse events (i.e., grade and frequency)
MTD of ibrutinib with anti-fungal prophylaxis when given with TEDD-R | after one cycle
  AEs will be tabulated and reported
MTD of ibrutinib when given with TEDD-R | after one cycle
  AEs will be tabulated and reported
Complete Response rate in untreated PCNSL patients | every 3 months for 1 year, every 4 months year 2, every 6 months year 3 then yearly
  The response rate will be determined and reported along with a 95% confidence interval

SECONDARY OUTCOMES:
Safety and Tolerability | Initiation of ibrutinib until 30 days after treatment
  Incidence of adverse events (i.e., grade and frequency)
Progression-free survival | every 3 months for 1 year, every 4 months year 2, every 6 months year 3 then yearly
  The response rate will be determined and reported along with a 95% confidence interval
Overall survival | every 3 months for 1 year, every 4 months year 2, every 6 months year 3 then yearly
  The response rate will be determined and reported along with a 95% confidence interval

CONTACTS AND LOCATIONS:
Overall Officials: Rahul Lakhotia, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. @@@@@@@@@@@@In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP. @@@@@@@@@@@@All collected IPD will be shared with collaborators under the terms of collaborative agreements.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data will be available during the study and indefinitely.@@@@@@@@@@@@Genomic data will be available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.@@@@@@Genomic data will be made available via dbGaP through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2014-C-0157.html